CLINICAL TRIAL: NCT00842205
Title: Role of Heme Oxygenase in the Pathogenesis od Hepatocellular Injury in Chronic HCV Infection
Brief Title: Role of Heme Oxygenase in the Pathogenesis of Hepatocellular Injury in Chronic Hepatitis C Virus (HCV) Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: IGA MZ, Czech Republic (Unknown)
Responsible Party: Petr Urbanek, Doc. MUDr., CSc, Dept of Internal Medicine, 1st Medical Faculty Charles University and Central Military Hospital Prague, Czech Republic
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IGA MZ CR NR9412-3
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Chronic HCV Infection; Nonalcoholic Steatohepatitis
Keywords: hepatitis C; NASH; Hem Oxygenase; Gene polymorphism
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hepatitis C | interventions — peginterferon alfa-2a; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 HCV positive pts (Active Comparator): Patients with chronic HCV infection undergoing liver biopsy followed by antiviral treatment.
  peg-IFN alfa 2a 180ug s.c. QW + ribavirin 1000-1200mg p.o. daily 48weeks or peg-IFN alfa 2b 1.5 ug/kg s.c. QW + ribavirin 100-1200mg p.o. daily 48 weeks
  Interventions: Drug: pegylated interferon; Drug: Ribavarin
- 2 Other liver disease (No Intervention): pts. with NASH (or other liver disease) undergoing liver biopsy.

INTERVENTIONS:
Drug: pegylated interferon — peg-IFN alfa 2a 180ug s.c. QW or peg-IFN alfa 2b 1.5 ug/kg s.c. QW
  Other Names: Pegasys; Pegintron
  Arms: 1 HCV positive pts
Drug: Ribavarin — ribavirin 1000-1200mg p.o. daily 48weeks or ribavirin 100-1200mg p.o. daily 48 weeks
  Other Names: Copegus; Rebetol
  Arms: 1 HCV positive pts

SUMMARY:
In the presented project, the role of heme oxygenase 1 and 2 in the procesess associated with fibroproduction in the chronic HCV infection will be studied. Heme oxygenase expression will be evaluated by the techniques of molecular genetics and immunohistochemistry, both in the liver tissue and in peripheral blood mononuclear cells. These parameters will be correlated with basic virological and clinical characteristics of the chronic HCV infection. The investigators' expected results may help in understanding the mechanisms of fibroproduction in chronic HVC infection and, therefore, contribute to explain individual differences in the development of chronic HCV infection.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) is a single stranded positive RNA virus belonging to the Flaviviridae family. HCV is a major cause of chronic hepatitis and progressive liver fibrosis leading to cirrhosis. Currently, the mechanisms responsible for hepatocellular injury are not fully understood. Oxidative damage has been hypothesized to play a role in HCV-induced liver disease, with reactive oxygen species (ROS), generated from HCV-infected hepatocytes and infiltrating immune cells. Persistence of recurrent hepatocellular injury leads to wound-healing process in which oxidative stress, inflammatory response mediated by immune cells and/or cytokines, and activation of hepatic stellate cells (HSCs) contribute to cascade of fibrogenesis. HCV can infect peripheral blood mononuclear cells (PBMC) of patients with chronic HCV infection . PBMC play key roles both in innate and adaptive antigen-specific immunity and they constitute critical components of the immune response.Heme oxygenase (HO) is the rate-limiting enzyme in the heme catabolic pathway. It cleaves pro-oxidant heme into equimolar amounts of carbon monoxide (CO), free iron, and biliverdin, which is rapidly metabolized to bilirubin by biliverdin reductase.The human HO-1 gene is located at chromosome 22q12 and a variable number of tandem repeat polymorphism (VNTR) was identified in the proximal promoter region. It is suggested that these highly polymorphic (GT)n repeats could alter the transcriptional activity. In recent years, enhanced HO enzymatic activity has been reported - probably through its formation of bioactive products - to possess antioxidant, cytoprotective, and neurotransmitter activity and to play a role in anti-inflammatory functions . AIMS: AIM 1.To characterize HO expression in liver biopsies in patients with chronic hepatitis C comparing to expression in patients with other types of hepatitis (esp. autoimmune) and to normal liver tissue. To investigate the relationship between HO expression and hepatitis C virus concentration, duration of infection, level of fibrosis and inflammation, ALT, AST activities, bilirubin levels, response to the standard treatment and a level of apoptosis. AIM 2. To characterize HO expression in PBMC in patients with chronic hepatitis C before, in the week 12 and after the standard treatment (PEG-IFN+RBV). To correlate HO expression in PBMC with viral concentration in sera and a response to the standard treatment.AIM 3. To investigate HO polymorphisms in patients with chronic hepatitis C. AIM 4. To investigate UGT1A1 28 polymorphism which is responsible for benign hyperbilirubinemia. Expected results: 1. This study could elucidate a relationship between development of liver fibrosis and inflammation and HO expression. 2. This project may, for the first time, show the relationship between chronic HCV infection and regulation of HO expression in PBMC. 3.This project will answer the question whether genetic predisposition, length polymorphism in HO promoter responsible for its lower transcriptional activity, could be a risk factor for fibrosis/cirrhosis development in patients infected with hepatitis C virus. UGT1A1 28 polymorphism is connected with low prevalence of diseases in which the oxidative stress is increased. We suggest that HCV infected persons might have low prevalence of this polymorphism or this polymorphism might be connected to low efficacy of antiviral treatment in these persons.

ELIGIBILITY:
Inclusion Criteria:

* chronic HCV infection
* must undergo liver biopsy
* must undergo antiviral treatment

Exclusion Criteria:

* liver sample not obtained
* blood samples for HCV testing not obtained in specified time points during antiviral therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
1. the relation between HO activity and basic virologic and histologic parameters in chronic HCV patients. 2. changes of HO activity within antiviral treatment 3. relation of HO gene polymorphisms to the course of disease | from HCV transmission in each individual patient to the time of liver biopsy and begining of antiviral treatment

SECONDARY OUTCOMES:
Relation of HO gene polymorphisms and UGT1A1*28 polymorphism. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cetral Military Hospital, Prague, Czechia

REFERENCES:
- [Derived] Urbanek P, Lenicek M, Muchova L, Subhanova I, Dusek L, Kasprikova N, Hrabal P, Bruha R, Vitek L. No association of promoter variations of HMOX1 and UGT1A1 genes with liver injury in chronic hepatitis C. Ann Hepatol. 2011 Oct-Dec;10(4):445-51. PMID 21911884